CLINICAL TRIAL: NCT00946491
Title: An Open-Label, Single-Dose, Crossover Study to Determine the Bioequivalency of Generic Haloperidol Tablets vs. Haldol in Normal Volunteers.
Brief Title: To Demonstrate the Relative Bioequivalency of Generic Haloperidol Tablets Versus Haldol in Normal Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D, VP of Product Development, Sandoz Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 87-01
Record Dates: First submitted 2009-07-24; First posted 2009-07-27 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2009-07

CONDITIONS: Psychosis
Keywords: Typical Antipsychotic
MeSH Terms: conditions — Psychotic Disorders | interventions — Haloperidol

ARMS (2):
- 1 (Experimental): Haloperidol 10 mg Tablets (Cord Laboratories)
  Interventions: Drug: Haloperidol 10 mg Tablets (Cord Laboratories)
- 2 (Active Comparator): Haldol 10 mg Tablets (McNeil Pharmaceuticals)
  Interventions: Drug: Haldol 10 mg Tablets (McNeil Pharmaceuticals)

INTERVENTIONS:
Drug: Haloperidol 10 mg Tablets (Cord Laboratories)
  Arms: 1
Drug: Haldol 10 mg Tablets (McNeil Pharmaceuticals)
  Arms: 2

SUMMARY:
To demonstrate the relative bioequivalency of generic Haloperidol tablets versus Haldol in normal volunteers.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal finding on physical exam, medical history, or clinical laboratory results on screening.

Exclusion Criteria:

* Positive test results for HIV or hepatitis B or C.
* Treatment for drug or alcohol dependence.

Ages: 35 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 1987-04; Primary Completion 1987-05 (Actual); Study Completion 1987-05 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on AUC and Cmax | 17 days

CONTACTS AND LOCATIONS:
Overall Officials: Philip T. Leese, M.D., Principal Investigator — Quincy Research Center